CLINICAL TRIAL: NCT04647968
Title: Primary vs Secondary Closure of Tracheo-cutaneous Fistulas: A Randomized Controlled Study
Brief Title: Primary vs Secondary Closure of Tracheo-cutaneous Fistulas
Acronym: TRACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Simon Brisebois, Assistant Professor - Division of Otolaryngology - Head & Neck Surgery, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-3699
Record Dates: First submitted 2020-11-12; First posted 2020-12-01 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Tracheostomy Complication; Post Tracheostomy Complications; Tracheostomy
Keywords: tracheostomy; tracheostomy closure; tracheocutaneous fistula

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: No masking because it is a surgical procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary closure of tracheo-cutaneous fistula (Other): This group will undergo a protocoled primary closure of their tracheotomy.
  Interventions: Procedure: Primary closure of tracheo-cutaneous fistula
- Secondary closure of tracheo-cutaneous fistula (Other): This group will undergo a protocoled secondary closure of their tracheotomy.
  Interventions: Procedure: Secondary closure of tracheo-cutaneous fistula

INTERVENTIONS:
Procedure: Primary closure of tracheo-cutaneous fistula — This procedure will follow protocoled steps. It consists of a sutured closure of the tracheotomy following local anesthesia, done at bedside.
  Arms: Primary closure of tracheo-cutaneous fistula
Procedure: Secondary closure of tracheo-cutaneous fistula — This procedure will follow protocoled steps. It consists of removing the tracheotomy canula and applying ointment and an Elastoplast on the site, which will be changed regularly until full healing of the wound.
  Arms: Secondary closure of tracheo-cutaneous fistula

SUMMARY:
The mean of this study is to compare primary and secondary closure of tracheo-cutaneous fistulas and evaluate the differences in outcomes between both techniques.

DETAILED DESCRIPTION:
In this study the investigators wish to recruit patients with a tracheotomy that has been installed for various reasons and that is ready for closure. The investigators intend to randomly allocate them a mean of closure, either primary or secondary. Once the fistula is closed, the investigators will follow them over a substantial period of time to compare outcomes of each mean of closing. Different questionnaires will be used to best evaluate a range of variables.

ELIGIBILITY:
Inclusion Criteria:

* Being covered by the RAMQ
* Having a tracheostomy either percutaneous or surgical
* Being ready for canula removal and closure of the fistula

Exclusion Criteria:

* Presenting a contraindication to primary tracheotomy closure (granuloma)
* Unable to consent
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction in regards to the scar (change) | 1 week, 1 month, 3 months, 6 months
  This outcome will evaluate patient satisfaction in regards to his tracheotomy scar following closure, measured with the Patient observer scar assesment scale (POSAS) validated questionnaire. A high score means a worse outcome.

SECONDARY OUTCOMES:
Healing time | 6 months
  This outcome will evaluate time until full closure of the wound using both methods of closure.
Respiratory complications | 6 months
  The investigators wish to establish whether there is a difference in respiratory complications occurence between the two means of closure.
Self reported quality of life related to dysphonia (change) | 1 week, 1 month, 3 months, 6 months
  The goal of this outcome is to evaluate the self reported quality of life of patients following tracheotomy closed by either mean. The investigators are going to use the Voice Handicap Index (VHI-10) validated questionnaire to better assess this outcome. A high score means a worse outcome, the highest score being 40.
Persisting fistula | 6 months
  This outcome intends to evaluate the frequency of persisting fistula using either method of closure.
Self reported quality of life related to dysphagia (change) | 1 week, 1 month, 3 months, 6 months
  The goal of this outcome is to evaluate the self reported quality of life of patients following tracheotomy closed by either mean. We are going to use the EAT-10 validated questionnaire to better assess this outcome. A high score means a worse outcome, the highest score being 40.
Self reported quality of life related to dyspnea (change) | 1 week, 1 month, 3 months, 6 months
  The goal of this outcome is to evaluate the self reported quality of life of patients following tracheotomy closed by either mean. This will be measure by the Dyspnea Index (DI) validated questionnaire but also with the follow-up history. The Dyspnea Index questionnaire has a maximum score of 40. A high score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brisebois, MD, MSC, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No